CLINICAL TRIAL: NCT06619392
Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics of HRS-2129 and the Food Effect on Pharmacokinetics Following Single Dose Administration in Healthy Subjects
Brief Title: A Single Dose Escalation Trial of HRS-2129 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-2129-101
Record Dates: First submitted 2024-09-23; First posted 2024-10-01 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: HRS-2129 for dose escalation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Treatment at dose level 1 (Experimental)
  Interventions: Drug: HRS-2129; Drug: HRS-2129 Placebo
- Treatment at dose level 2 (Experimental)
  Interventions: Drug: HRS-2129; Drug: HRS-2129 Placebo
- Treatment at dose level 3 (Experimental)
  Interventions: Drug: HRS-2129; Drug: HRS-2129 Placebo
- Treatment at dose level 4 (Experimental)
  Interventions: Drug: HRS-2129; Drug: HRS-2129 Placebo
- Treatment at dose level 5 (Experimental)
  Interventions: Drug: HRS-2129; Drug: HRS-2129 Placebo

INTERVENTIONS:
Drug: HRS-2129 — HRS-2129
Drug: HRS-2129 Placebo — HRS-2129 Placebo

SUMMARY:
The study is being conducted to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics in healthy subjects, and to evaluate the food effect on pharmacokinetics of HRS-2129.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 55 years old (inclusive);
2. Body weight: ≥ 50 kg for male and ≥ 45 kg for female, body mass index: 19.0 ~ 28.0 kg/m2 (inclusive);
3. Subject has no plan to give a birth, donate sperm or eggs from signing the informed consent form to 6 months after last dose;
4. Female subjects: non-pregnant or non-lactating;
5. The skin to receive pain stimuli has no wound or derma disease.
6. Subject who is willing to accept cold pain test.
7. Subject who voluntarily signs the informed consent.

Exclusion Criteria:

1. Subject who suffers from clinical acute and chronic diseases of circulatory system, endocrine system, nervous system, digestive system, respiratory system, hematology, immunology, psychiatry and metabolic abnormalities;
2. Subject with the following abnormalities: aspartate aminotransferase, alanine aminotransferase, total bilirubin, or serum creatine value exceeds the upper limit of the normal range, QTcF > 450 ms, hyperpotassemia or hypopotassemia;
3. Subject with a history of torsade de pointes, symptomatic ventricular arrhythmia, or personal or family history of short QT syndrome or long QT syndrome;
4. Subject with a history of allergies to the IMP or its excipients, or subject with allergic constitution;
5. Subject who underwent major surgery within 6 months prior to screening, or received surgery that may significantly affect the pharmacokinetics or safety evaluation of the IMP, or who plans to undergo surgery during the study period;
6. Subject with a medication history that inhibits or induces liver metabolism of drug has been used within 1 month before administration;
7. Subject with vaccinated within 1 month prior to screening or plan to be vaccinated during the study;
8. Subject who used any drugs or health products (including Chinese herbal medicines) within 7 half-lives or 14 days (whichever is longer) before administration, or who plans to receive other drug treatments during the study;
9. Subject who has participated in clinical trials and received experimental drugs within 3 months before screening, or plans to participate in other clinical trials during this study;
10. Donate blood/blood loss ≥ 400 mL within 3 months before screening;
11. Subject who smoked more than 5 cigarettes per day on average within 3 months before screening;
12. Drink more than 14 units of alcohol per week on average;
13. Drink excessive tea, coffee or caffeinated beverages within 3 months before screening;
14. Consume special food (such as grapefruit, grapefruit juice or food/drink containing grapefruit juice, chocolate, tobacco, alcohol, caffeine and other food or drink) within 48 hours before administration;
15. Subject who has special requirements for diet and cannot follow a unified diet;
16. Subject with clinical significant abnormalities in medical examination;
17. Subject with positive tests for hepatitis B surface antigen, hepatitis C virus antibody, syphilis or human immunodeficiency virus antibody;
18. Subject with a history of drug abuse or with a positive result for drug abuse test;
19. Alcohol test result is positive;
20. Subject who has difficulty in swallowing, or venous blood collection, or who cannot tolerate venipuncture, or who has a history of fainting of needle or blood;
21. Subject may not be able to complete the study due to other reasons or the investigators considers that he is not suitable for inclusion.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2024-10-17 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
The incidence and severity of adverse events | from ICF signing date to day 28 since last dose

SECONDARY OUTCOMES:
Pharmacokinetic parameter of HRS-2129: Cmax | 0 hour to 216 hour after administration
Pharmacokinetic parameter of HRS-2129: AUC0-t | 0 hour to 216 hour after administration
Pharmacokinetic parameter of HRS-2129: AUC0-inf | 0 hour to 216 hour after administration
Pharmacokinetic parameter of HRS-2129: Tmax | 0 hour to 216 hour after administration
Pharmacokinetic parameter of HRS-2129: t1/2 | 0 hour to 216 hour after administration
Pharmacokinetic parameter of HRS-2129: CL/F | 0 hour to 216 hour after administration
Pharmacokinetic parameter of HRS-2129: Vz/F | 0 hour to 216 hour after administration
Electrocardiogram measurement: QTcF interval | 90 minute predose to 48 hour after administration
Pain detection threshold for the Thermode Cold Test | 0 hour to 12 hour after administration
Pain tolerance time for the Thermode Cold Test | 0 hour to 12 hour after administration

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided